CLINICAL TRIAL: NCT04034836
Title: Parecoxib as an Adjuvant to Scalp Nerve Blocks for Relief of Post-craniotomy Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY 2018-034-02-2
Record Dates: First submitted 2019-07-21; First posted 2019-07-26 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Pain, Postoperative; Neurosurgery
Keywords: Pain, Postoperative; Parecoxib; Ropivacaine; Scalp nerve blocks; Craniotomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; parecoxib

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The scalp blocks group (Experimental): The scalp blocks group will receive scalp blocks with ropivacaine, 20ml, plus 10 mg parecoxib (diluted in 2 mL NS) with epinephrine (5 ug/mL) and i.v. saline 2ml;
  Interventions: Drug: Scalp blocks with ropivacaine plus parecoxib
- The i.v. group (Active Comparator): The i.v. group will receive scalp blocks with ropivacaine 20ml, plus saline 2ml with epinephrine (5 ug/mL) together with 10 mg parecoxib (diluted in 2 mL NS) intravenously.
  Interventions: Drug: Scalp blocks with ropivacaine and intravenous parecoxib
- The control group (Active Comparator): The control group will receive scalp blocks with ropivacaine, 20ml, plus saline 2ml with epinephrine (5 ug/mL) and i.v. saline 2ml;
  Interventions: Drug: Scalp blocks with ropivacaine and intravenous saline

INTERVENTIONS:
Drug: Scalp blocks with ropivacaine plus parecoxib — Scalp blocks with ropivacaine 0.75% wt/vol, 20ml, plus 10 mg parecoxib (diluted in 2 mL NS) with epinephrine at 1:200,000 (5 ug/mL) and i.v. saline 2ml;An independent researcher will prepare the study solution in a separate operating room. The study solutions with syringes (50-ml) for the scalp blocks and syringes (5-ml) for intravenous injection are prepared and numbered with a 23-gauge needle by an independent researcher, after opening the envelope containing the allocation of treatment. After induction, the assigned solutions will be injected subcutaneously or intravenously separately by the anesthesiologist. The scalp blocks will be performed along the lines of the technique previously described by Pinosky et al. The following nerves were blocked bilaterally: the supraorbital and supratrochlear nerves; the zygomatico-temporal nerves; the auriculotemporal nerves; the postauricular branches of the greater auricular nerves; the greater, lesser, and third occipital nerves.
  Arms: The scalp blocks group
Drug: Scalp blocks with ropivacaine and intravenous parecoxib — Scalp blocks with ropivacaine 0.75% wt/vol, 20ml, plus saline 2ml with epinephrine at 1:200,000 (5 ug/mL) together with 10 mg parecoxib (diluted in 2 mL NS) intravenously. An independent researcher will prepare the study solution in a separate operating room. The study solutions with syringes (50-ml) for the scalp blocks and syringes (5-ml) for intravenous injection are prepared and numbered with a 23-gauge needle, after opening the envelope containing the allocation of treatment. After induction, the assigned solutions will be injected subcutaneously or intravenously separately by the anesthesiologist. The scalp blocks will be performed along the lines of the technique previously described by Pinosky et al. The following nerves were blocked bilaterally: the supraorbital and supratrochlear nerves; the zygomatico-temporal nerves; the auriculotemporal nerves; the postauricular branches of the greater auricular nerves; the greater, lesser, and third occipital nerves.
  Arms: The i.v. group
Drug: Scalp blocks with ropivacaine and intravenous saline — Scalp blocks with ropivacaine 0.75% wt/vol, 20ml, plus saline 2ml with epinephrine at 1:200,000 (5 ug/mL) and i.v. saline 2ml. An independent researcher will prepare the study solution in a separate operating room. The study solutions with syringes (50-ml) for the scalp blocks and syringes (5-ml) for intravenous injection are prepared and numbered with a 23-gauge needle by an independent researcher, after opening the envelope containing the allocation of treatment. After induction, the assigned solutions will be injected subcutaneously or intravenously separately by the anesthesiologist. The scalp blocks will be performed along the lines of the technique previously described by Pinosky et al. The following nerves were blocked bilaterally: the supraorbital and supratrochlear nerves; the zygomatico-temporal nerves; the auriculotemporal nerves; the postauricular branches of the greater auricular nerves; the greater, lesser, and third occipital nerves.
  Arms: The control group

SUMMARY:
Pain is common for the first 2 days after major craniotomy. Inadequate analgesia induced sympathetically mediated hypertension may lead to an increased risk for post-operative complications, such as arterial hypertension, intracranial hemorrhage, prolonged hospital stay, and mortality.Pain after craniotomy derives from the scalp and pericranial muscles.Scalp block with local anesthesia seems to provide effective and safe anesthetic management.Scalp block can be performed by directly blocking the six different nerves that provide the sensory innervation of the scalp in neurological surgery.Even if adrenaline as an additive agent, scalp block using 0.5% or 0.75% bupivacaine with adrenaline could only improve postoperative analgesic for up to six hours after craniotomy.However, pain is common for the first 2 days after major elective intracranial surgery, and the relatively short analgesic time of scalp nerve blocks does not seem to meet the requirements of craniotomy. Therefore, how to improve the quality and duration of scalp nerve blocks with local anesthetics is of great significance.Parecoxib is a NSAIDs that specifically inhibits the enzyme COX-2.Liu et al firstly applied parecoxib as an adjuvant to local anesthetics on peripheral nerve blocks and reported 20 mg parecoxib added to ropivacaine injected locally on the brachial plexus nerve prolonged the motor and sensory block times of the nerve blockade and ameliorated postoperative pain intensity for patients receiving forearm orthopaedic surgery. However, there has not been reported about local application of parecoxib on scalp nerve blocks. The investigators postulate that parecoxib may be also ideal for scalp nerve blocks for relief of post-craniotomy pain, and further research is needed.

The APONIA trial aims to establish whether scalp blocks with a mixture of ropivacaine plus parecoxib is able to relieve patients' postoperative pain compared with local anesthetics alone, thereby potentially changing medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 64 years
* American Society of Anesthesiologists (ASA) physical status of I, II and III
* Preoperative Glasgow Coma Scale (GCS) score of 15/15
* Scheduled for elective craniotomy under general anesthesia

Exclusion Criteria:

* Patients with chronic headache or chronic pain syndrome for any reason
* Patients with psychiatric disorders, uncontrolled epilepsy, coagulopathy, infection around puncture point
* Inability to understand and incapacity to use the pain scales before surgery
* Pregnancy or at breastfeeding;
* Participation in another intervention trial that interferes with the intervention or outcome of this trial
* History of allergies to any of the study drugs
* Refusal to participate or unable to acquire informed consent provided by the patients and/or legal guardian
* Having their first craniotomy surgery with an occipital bone defect
* Excessive alcohol or drug abuse, chronic opioid use (more than 2 weeks or 3 days per week for more than 1 month), use of drugs with confirmed or suspected sedative or analgesic effects, use of any painkiller within 24 hours before surgery
* Extreme body mass index (BMI) (< 15 or > 35);

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-10-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The time to the first rescue analgesic | Within 48 hours after the operation
  Postoperatively, when the patient reports an NRS score of 4 or more or at the request of the patient, patients will be treated with morphine 2 mg intravenously as first rescue analgesic. Morphine 5 mg intravenously will be used as a second rescue analgesic if the NRS remained at 4 despite the use of morphine 2 mg.

SECONDARY OUTCOMES:
Numerical rating scale of pain | At 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 20 hours, 24 hours, 48 hours after surgery
  Pain will be assessed after surgery by a numerical rating scale (0 indicates no pain, 10 indicates the most severe pain imaginable)
Glasgow Coma Scale (GCS) score | At 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 20 hours, 24 hours, 48 hours after surgery
  The scale is composed of three tests: eye, verbal and motor responses. The three values separately as well as their sum are considered. The lowest possible GCS (graded 1 in each element) is 3 (deep coma or death), while the highest is 15 (fully awake person).
The doses of extra sufentanil boluses | During the surgery
  Intraoperative analgesic requirement defined as extra sufentanil boluses required to blunt significant sympathetic response to surgical stimulation will be recorded.
Number of participates using extra sufentanil boluses | During the surgery
  Intraoperative analgesic requirement defined as extra sufentanil boluses required to blunt significant sympathetic response to surgical stimulation will be recorded.
Number of participates with postoperative nausea and vomiting (PONV) | Within 48 hours postoperatively
  Vomiting will be defined as the forceful expulsion of gastric contents, and nausea will be defined as an unpleasant sensation associated with the urge to vomit.
Number of participates with bradycardia | Within 48 hours postoperatively
  An above 20% of decrease in heart rate from baseline values will be considered as clinically significant.
Number of participates with hypotension | Within 48 hours postoperatively
  An above 20% of decrease in blood pressure from baseline values will be considered as clinically significant
The time during PACU | Approximately 2 hours after the surgery
  Patients will be transferred to the postoperative care unit (PACU) after extubation. A modified Aldrete score > 9 will be required for discharge from the PACU to a ward. The time during PACU is defined as the duration in the PACU after surgery
Length of stay (LOS) | Approximately 2 weeks after the surgery
  LOS is defined as the number of nights spent in the hospital after surgery
Adverse Events | Approximately 2 weeks after the surgery
  An AE will be defined as any untoward medical occurrence, such as local hematoma, nerve injury, intra-arterial injection, allergic or toxic reaction, deriving facial nerve paralysis from scalp block.
Serious adverse events (SAEs) | Approximately 2 weeks after the surgery
  Serious adverse events (SAEs) will include death, immediately life-threatening conditions, coma, inpatient hospitalization or prolongation of existing hospitalization, et al.
patient satisfaction score (PSS) | At 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 20 hours, 24 hours, 48 hours after surgery
  Patient satisfaction will be assessed by the patient satisfaction score (PSS) (0 for unsatisfactory and 10 for very satisfactory)

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gottschalk A, Berkow LC, Stevens RD, Mirski M, Thompson RE, White ED, Weingart JD, Long DM, Yaster M. Prospective evaluation of pain and analgesic use following major elective intracranial surgery. J Neurosurg. 2007 Feb;106(2):210-6. doi: 10.3171/jns.2007.106.2.210. PMID 17410701
- [Background] Basali A, Mascha EJ, Kalfas I, Schubert A. Relation between perioperative hypertension and intracranial hemorrhage after craniotomy. Anesthesiology. 2000 Jul;93(1):48-54. doi: 10.1097/00000542-200007000-00012. PMID 10861145
- [Background] Flexman AM, Ng JL, Gelb AW. Acute and chronic pain following craniotomy. Curr Opin Anaesthesiol. 2010 Oct;23(5):551-7. doi: 10.1097/ACO.0b013e32833e15b9. PMID 20717011
- [Background] Dunn LK, Naik BI, Nemergut EC, Durieux ME. Post-Craniotomy Pain Management: Beyond Opioids. Curr Neurol Neurosci Rep. 2016 Oct;16(10):93. doi: 10.1007/s11910-016-0693-y. PMID 27604271
- [Background] Chaki T, Sugino S, Janicki PK, Ishioka Y, Hatakeyama Y, Hayase T, Kaneuchi-Yamashita M, Kohri N, Yamakage M. Efficacy and Safety of a Lidocaine and Ropivacaine Mixture for Scalp Nerve Block and Local Infiltration Anesthesia in Patients Undergoing Awake Craniotomy. J Neurosurg Anesthesiol. 2016 Jan;28(1):1-5. doi: 10.1097/ANA.0000000000000149. PMID 25493926
- [Background] Lee EJ, Lee MY, Shyr MH, Cheng JT, Toung TJ, Mirski MA, Chen TY. Adjuvant bupivacaine scalp block facilitates stabilization of hemodynamics in patients undergoing craniotomy with general anesthesia: a preliminary report. J Clin Anesth. 2006 Nov;18(7):490-4. doi: 10.1016/j.jclinane.2006.02.014. PMID 17126775
- [Background] Nguyen A, Girard F, Boudreault D, Fugere F, Ruel M, Moumdjian R, Bouthilier A, Caron JL, Bojanowski MW, Girard DC. Scalp nerve blocks decrease the severity of pain after craniotomy. Anesth Analg. 2001 Nov;93(5):1272-6. doi: 10.1097/00000539-200111000-00048. PMID 11682413
- [Background] Bala I, Gupta B, Bhardwaj N, Ghai B, Khosla VK. Effect of scalp block on postoperative pain relief in craniotomy patients. Anaesth Intensive Care. 2006 Apr;34(2):224-7. doi: 10.1177/0310057X0603400203. PMID 16617645
- [Background] Romsing J, Moiniche S. A systematic review of COX-2 inhibitors compared with traditional NSAIDs, or different COX-2 inhibitors for post-operative pain. Acta Anaesthesiol Scand. 2004 May;48(5):525-46. doi: 10.1111/j.0001-5172.2004.00379.x. PMID 15101847
- [Background] Romsing J, Moiniche S, Ostergaard D, Dahl JB. Local infiltration with NSAIDs for postoperative analgesia: evidence for a peripheral analgesic action. Acta Anaesthesiol Scand. 2000 Jul;44(6):672-83. doi: 10.1034/j.1399-6576.2000.440607.x. PMID 10903014
- [Background] Koppert W, Wehrfritz A, Korber N, Sittl R, Albrecht S, Schuttler J, Schmelz M. The cyclooxygenase isozyme inhibitors parecoxib and paracetamol reduce central hyperalgesia in humans. Pain. 2004 Mar;108(1-2):148-53. doi: 10.1016/j.pain.2003.12.017. PMID 15109518
- [Background] Williams DL, Pemberton E, Leslie K. Effect of intravenous parecoxib on post-craniotomy pain. Br J Anaesth. 2011 Sep;107(3):398-403. doi: 10.1093/bja/aer223. PMID 21841050
- [Background] Liu X, Zhao X, Lou J, Wang Y, Shen X. Parecoxib added to ropivacaine prolongs duration of axillary brachial plexus blockade and relieves postoperative pain. Clin Orthop Relat Res. 2013 Feb;471(2):562-8. doi: 10.1007/s11999-012-2691-y. Epub 2012 Nov 21. PMID 23179117
- [Background] Krauss P, Marahori NA, Oertel MF, Barth F, Stieglitz LH. Better Hemodynamics and Less Antihypertensive Medication: Comparison of Scalp Block and Local Infiltration Anesthesia for Skull-Pin Placement in Awake Deep Brain Stimulation Surgery. World Neurosurg. 2018 Dec;120:e991-e999. doi: 10.1016/j.wneu.2018.08.210. Epub 2018 Sep 7. PMID 30196173